CLINICAL TRIAL: NCT05948670
Title: An Exploratory Randomized Controlled Trial of Participant Satisfaction With the BUILD Mobile Application
Brief Title: Participant Satisfaction With the BUILD Mobile Application
Status: Completed | Phase: Not Applicable | Type: Interventional
Sponsor: Woebot Health (Industry)
Responsible Party: Sponsor
Allocation: Randomized | Model: Parallel | Masking: Double | Purpose: Other
Other Study IDs: W-DISC-001
Record Dates: First submitted 2023-06-23; First posted 2023-07-17 (Actual); Results first posted 2025-01-07 (Actual); Last update posted 2025-02-18 (Actual); Status verified 2025-01

CONDITIONS: Satisfaction, Personal
Keywords: Woebot; LLM; Relational agent
MeSH Terms: conditions — Personal Satisfaction

STUDY DESIGN:
Intervention Model Description: 1:1 randomization
Who Masked: Participant, Investigator
Oversight: Data Monitoring Committee: No | FDA-regulated Drug: No | FDA-regulated Device: Yes | Unapproved Device: Yes | US Export: No

ARMS (2):
- DISC-MVP (Experimental): Participants randomized to the experimental condition, DISC-MVP, will be asked to download and use the BUILD study application. They will have access to the app throughout the 2 week study.
  Interventions: Device: DISC-MVP
- DISC-CON (Active Comparator): Participants randomized to the digital control condition, DISC-CON, will be asked to download and use the BUILD study application. They will have access to the app throughout the 2 week study.
  Interventions: Device: DISC-CON

INTERVENTIONS:
Device: DISC-MVP — DISC-MVP is a digital program grounded in validated psychotherapies (e.g., cognitive behavioral therapy), that enlists a relational agent (Woebot) to engage users in therapeutic conversations and generates responses through a controlled process using large language models.
  Arms: DISC-MVP
Device: DISC-CON — DISC-CON is a digital program grounded in validated psychotherapies (e.g., including cognitive behavioral therapy) that uses a virtual relational agent (Woebot) to engage users in therapeutic conversations with responses that are selected from a list based on natural language processing.
  Arms: DISC-CON

SUMMARY:
This study explores user satisfaction with the BUILD mobile application.

DETAILED DESCRIPTION:
This exploratory randomized, double-blind, controlled trial explores user satisfaction with the BUILD mobile application. The BUILD app uses a relational agent (Woebot) to engage users in therapeutic conversations. Eligible participants will be randomized to one of two treatment conditions: (1) an experimental condition in which Woebot uses large language models to understand user sentiment, and based on this understanding of natural language generate responses through a controlled process or (2) a digital control condition in which Woebot selects from a list of responses based on natural language processing. Participants will receive instructions on downloading and using the BUILD app in order to access the intervention to which they were assigned. Participants will use the app as instructed and will complete assessments for the primary endpoint at Week 2 (EOT) with additional measures being collected at Baseline, Day 3, and Week 2. Results from this study will provide preliminary data on user satisfaction and feasibility and inform product development iteration for inclusion in a statistically powered clinical randomized controlled trial.

ELIGIBILITY:
Inclusion Criteria:

1. Must be 18+ years of age and older
2. Must own or have regular access to a smartphone with a recent operating system installed (Android: OS 8.0 or higher, Apple: iOS 13.0 or higher) with reliable Wi-Fi access or sufficient data plan to engage with assigned treatment condition for the duration of the study
3. Must be available and committed to engage with the program and complete assessments for a 2-week duration
4. Must be able to read and write in English
5. Must have primary residence in the United States

Exclusion Criteria:

1. Current suicidal ideation with a plan and/or intent or a suicide attempt within the past 12 months
2. Previous Woebot use

Min Age: 18 Years | Sex: All | Healthy Volunteers: Yes
Age Groups: Adult, Older Adult
Enrollment: 175 (Actual)
Dates: Start 2023-10-04 (Actual); Primary Completion 2023-11-15 (Actual); Study Completion 2023-11-15 (Actual)

CONTACTS AND LOCATIONS:
Overall Officials: Tim Campellone, PhD, Principal Investigator — Woebot Health
Locations (1):
- Woebot Investigational Site, San Francisco, California, United States

REFERENCES:
- [Derived] Campellone TR, Flom M, Montgomery RM, Bullard L, Pirner MC, Pavez A, Morales M, Harper D, Oddy C, O'Connor T, Daniels J, Eaneff S, Forman-Hoffman VL, Sackett C, Darcy A. Safety and User Experience of a Generative Artificial Intelligence Digital Mental Health Intervention: Exploratory Randomized Controlled Trial. J Med Internet Res. 2025 May 23;27:e67365. doi: 10.2196/67365. PMID 40408143

RESULTS

PARTICIPANT FLOW:
Period: Overall Study
Arm/Group | DISC-MVP | DISC-CON
Started | 87 | 88
Completed | 81 | 79
Not Completed | 6 | 9
Not completed — Protocol Violation | 6 | 8
Not completed — Withdrawal by Subject | 0 | 1

BASELINE CHARACTERISTICS:
Groups:
- Total: Total of all reporting groups
Arm/Group | DISC-MVP | DISC-CON | Total
Number analyzed (Participants) | 81 | 79 | 160
Age, Continuous [Mean (Standard Deviation); unit: years] | 41.99 (12.85) | 45.70 (15.09) | 43.82 (14.08)
Sex: Female, Male [Count of Participants; unit: Participants]
  Female | 57 | 60 | 117
  Male | 24 | 19 | 43
Ethnicity (NIH/OMB) [Count of Participants; unit: Participants]
  Hispanic or Latino | 9 | 8 | 17
  Not Hispanic or Latino | 72 | 71 | 143
  Unknown or Not Reported | 0 | 0 | 0
Race (NIH/OMB) [Count of Participants; unit: Participants]
  American Indian or Alaska Native | 0 | 2 | 2
  Asian | 5 | 3 | 8
  Native Hawaiian or Other Pacific Islander | 0 | 0 | 0
  Black or African American | 22 | 25 | 47
  White | 47 | 47 | 94
  More than one race | 5 | 0 | 5
  Unknown or Not Reported | 2 | 2 | 4
Region of Enrollment [Number; unit: participants]
  United States | 81 | 79 | 160

OUTCOME MEASURES:

1. Primary Outcome: User Satisfaction as Measured by the Client Satisfaction Questionnaire (CSQ-8)
Description: The CSQ-8 is an 8-item measure used to assess client's satisfaction with treatment.Total scores range from 8-32, with high scores indicating greater satisfaction with the treatment.
Time Frame: Post-intervention at Week 2
Measure: Mean (Standard Deviation); unit: score on a scale
Arm/Group | DISC-MVP | DISC-CON
Number analyzed (Participants) | 81 | 79
score on a scale | 23.49 (6.30) | 23.97 (5.95)

2. Secondary Outcome: User Satisfaction Amongst a Sub-sample of Adults With at Least Mild Symptoms of Depression and/or Anxiety.
Description: as for outcome 1
Time Frame: Post-intervention at Week 2
Measure: Mean (Standard Deviation); unit: score on a scale
Arm/Group | DISC-MVP | DISC-CON
Number analyzed (Participants) | 66 | 62
score on a scale | 22.95 (6.49) | 23.68 (6.03)

ADVERSE EVENTS:
Time Frame: 2 weeks
Arm/Group | DISC-MVP | DISC-CON
All-Cause Mortality (participants affected / at risk) | 0/87 | 0/88
Serious Adverse Events (participants affected / at risk) | 0/87 | 0/88
Other Adverse Events (participants affected / at risk) | 1/87 | 7/88
OTHER ADVERSE EVENTS; cells are participants affected of the arm's N at risk (number of events):
Term (organ system) | DISC-MVP (N=87) | DISC-CON (N=88)
Worsening physical health condition (General disorders) | 0 (0) | 2 (2)
Worsening mental health condition (Psychiatric disorders) | 0 (0) | 3 (3)
New physical health condition (General disorders) | 1 (1) | 2 (2)

CERTAIN AGREEMENTS:
Principal investigators are sponsor employees: Yes

DOCUMENTS (1):
  • Study Protocol and Statistical Analysis Plan (2023-09-08): https://cdn.clinicaltrials.gov/large-docs/70/NCT05948670/Prot_SAP_000.pdf